CLINICAL TRIAL: NCT01099371
Title: Progressive Resistance Training in Women With Knee Osteoarthritis
Brief Title: Resistance Training in Knee Osteoarthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Renata Trajano Borges e Jorge, Federal University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDAAAA
Record Dates: First submitted 2010-04-01; First posted 2010-04-07 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2009-01

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise (Experimental)
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — progressive resistance training

SUMMARY:
The purpose of this study is to determine whether:

1. Progressive resistance training improves pain and disability
2. Progressive Resistance training improves muscular strength, ability to walk and quality of life

DETAILED DESCRIPTION:
Patients in experimental group participated in a 12-week progressive resistance training using a repetition maximum (RM) exercise in which patients performed 1RM with the maximum bearable weight. Once the 1RM was determined, training was divided into the following regimen: 2 series of 8 repetitions, the first with 50% and the second with 70% of 1RM.

The exercises were knee extension and flexion and hip abduction and adduction, all performed in machines. The 1RM load was reevaluated every 2 weeks.

The control group remained on a three-month waiting list for physiotherapy. Patients were assessed for pain, function, quality of life, muscle strength and six-minute walk test.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Age between 40-70 years old
* Pain between 3 and 8 on a 10-point numeric pain scale
* Radiographically confirmed knee OA

Exclusion Criteria:

* Inflammatory diseases or any comorbidity that prohibit exercises, regular physical activity
* Trip plans for the next 12 months

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Pain assessed on a 10-point numeric pain scale | week 0
  Scale: visual analog scale

SECONDARY OUTCOMES:
Disability assessed on WOMAC | week 6
  Western Ontario McMaster University Osteoarthritis Index Rheumatology An arthritic pain scoring system ranging from 0-no pain/disability to 100-most severe pain/disability
  WOMAC-pain, WOMAC-function and WOMAC-stifness
Quality of life assessed on the SF-36 | week 6
  Questionnaire Short-form-36
Six-minute walk test | week 12
  To assess distance walked in 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Natour, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil